CLINICAL TRIAL: NCT01353079
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Group Efficacy And Safety Trial Of Sublingual-Oral Immunotherapy (SLIT) In Adults With Allergic Rhinoconjunctivitis Caused By Ragweed Pollen
Brief Title: Efficacy and Safety Study Of Short Ragweed Pollen Sublingual-Oral Immunotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Greer Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLIT10-01
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Results first posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-01

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short Ragweed Pollen Allergenic Extract (Experimental)
  Interventions: Biological: Short Ragweed Pollen Allergenic Extract
- Glycero-COCAs (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Short Ragweed Pollen Allergenic Extract — Daily sublingual administration of Short Ragweed Pollen Allergenic Extract up to 42 U Amb a 1 for a minimum of 8 weeks prior to the ragweed pollen season.
  Arms: Short Ragweed Pollen Allergenic Extract
Biological: Placebo — Placebo: Glycero-COCAs sublingual
  Arms: Glycero-COCAs

SUMMARY:
The primary objective of this study is to demonstrate that SLIT administered pre-and co-seasonally is effective in reducing rhinoconjunctivitis symptoms during the entire short ragweed pollen season.

ELIGIBILITY:
Inclusion Criteria:

* allergic to ragweed

Exclusion Criteria:

* not allergic to ragweed
* history of anaphylaxis
* subject with chronic sinusitis, unstable angina, significant arrhythmia, uncontrolled hypertension, or other chronic or immunological disease
* Asthmatic subjects with FEV1 or PEF less than or equal to 80% predicted
* Subjects who have received experimental drug within 30 days prior to study admission
* Subjects who have received anit-IgE medications in the last 12 months
* Subjects who have received ragweed immunotherapy in the last 3 years
* Subjects who are currently users of inhaled, intramuscular, or intravenous corticosteroids, tricyclic anti-depressants, beta blockers, and MAO inhibitors
* Subjects refusing to sign epi-pen training form
* Females who are pregnant or breast feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 429 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 7, Warrenton, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Short Ragweed Pollen Allergenic Extract: Allergy Immunotherapy: Daily administration of Ragweed Allergenic Extract up to 42 U Amb a 1 for a minimum of 8 week prior to the ragweed pollen season.
  Short Ragweed Allergenic Extract: Active-Short Ragweed Allergenic Extract sublingual
- Glycero-COCAs: Placebo-Glycero-COCAs sublingual
Period: Overall Study
Arm/Group | Short Ragweed Pollen Allergenic Extract | Glycero-COCAs
Started | 218 | 211
Completed | 191 | 190
Not Completed | 27 | 21

BASELINE CHARACTERISTICS:
Groups:
- Ragweed Allergenic Extract: Allergy Immunotherapy: Daily administration of Ragweed Allergenic Extract up to 42 U Amb a 1 for a minimum of 8 weeks prior to the ragweed pollen season.
  Short Ragweed Allergenic Extract: Active-Short Ragweed Allergenic Extract sublingual
- Glycero-COCAs: Placebo: Glycero-COCAS sublingual
- Total: Total of all reporting groups
Arm/Group | Ragweed Allergenic Extract | Glycero-COCAs | Total
Number analyzed (Participants) | 218 | 211 | 429
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 218 | 211 | 429
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 117 | 244
  Male | 91 | 94 | 185

OUTCOME MEASURES:

1. Primary Outcome: Scores on a Scale [Net Average Combined Daily Rhinoconjunctivitis Symptom (RSS) and Medication Scores]
Description: Change in baseline in avg combined daily RSS and medication scores during entire ragweed season in ITT population. Symptom score: sum of scores from 8 symptoms rated 0-3 (0=absent, 1=mild, 2=moderate, 3=severe), ocular (itchiness, swelling/redness, and watery eyes/tears), nasal (sneezing, itching, runny and stuffy nose), and ears (itching). Avg daily RSS computed by: (1) summing 8 individual allergy symptoms recorded in AM and PM; (2) forming daily RSS by summing AM and PM RSS for each day of ragweed season; (3) averaging daily RSS for entire ragweed season.Total allergy relief medication score computed by summing individual medication scores. Relief medication scores: 0-no medication taken; 1-using once daily oral antihistamine; 1-using once daily ocular antihistamine; 1-treatment with albuterol. Maximum medication score dependent on cumulative rescue medication use. Lower result is more favorable. Avg daily Combined Score Range: 0 (min) - 51 (max); lower score was more favorable.
Time Frame: 2011 ragweed pollen season, 8/2011 -10/2011
Population: ITT population includes subjects who had at least one post treatment efficacy measurement
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Ragweed Allergenic Extract: Allergy Immunotherapy: Daily sublingual administration of ragweed allergenic extract up to 42 U Amb a 1 for a minimum of 8 weeks prior to the ragweed pollen season.
  Short Ragweed Allergenic Extract: Active-Short Ragweed Allergenic Extract sublingual
- Placebo (Glycero-Cocas): Placebo: Glycero-COCAs sublingual
Arm/Group | Ragweed Allergenic Extract | Placebo (Glycero-Cocas)
Number analyzed (Participants) | 196 | 193
Scores on a scale | 0.853 (1.64) | 1.687 (2.40)
Statistical Analysis 1: Comparison: Ragweed Allergenic Extract vs Placebo (Glycero-Cocas); Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = -0.834, 95% CI 2-sided [-1.298 to -0.369]

2. Secondary Outcome: Scores on a Scale (Net Average Combined Daily Rhinoconjunctivitis Symptom and Medication Scores Reported During the Three Peak Weeks of Ragweed Pollen Season)
Description: Symptom score: sum of scores from 8 symptoms rated 0-3 (0=absent, 1=mild, 2=moderate, 3=severe), ocular (itchiness, swelling/redness, watery eyes/tears), nasal (sneezing, itching, runny, stuffy nose), and ears (itching). Avg daily RSS computed by summing 8 individual allergy symptoms recorded in AM and PM; forming daily RSS by summing AM and PM RSS for each day; averaging daily RSS for three peak weeks. Total allergy relief medication score computed by summing individual medication scores. Relief medication scores: 0-no medication taken; 1-using once daily oral antihistamine; 1-using once daily ocular antihistamine; 1-treatment with albuterol. Max medication score dependent on cumulative rescue medication use. Lower result, more favorable. Three peak weeks of ragweed pollen counts during entire ragweed season was contiguous and calculated using a moving average of ragweed pollen counts for each week. Avg daily Combined Score Range: 0 (min) - 51 (max); lower score was more favorable.
Time Frame: 3 peak weeks of the 2011 ragweed pollen season
Population: ITT population includes subjects who had at least one post treatment efficacy measurement. This analysis includes subjects the met the ITT criteria excluding those subjects that did not have either a combined symptom/medication score or RSS during the three peak weeks of the ragweed pollen season.
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Ragweed Allergenic Extract: Allergy Immunotherapy: Daily sublingual administration of Short Ragweed Allergenic Extract up to 42 U Amb a 1 for a minimum of 8 weeks prior to the ragweed pollen season.
  Short Ragweed Allergenic Extract: Active-Short Ragweed Allergenic Extract sublingual
Arm/Group | Ragweed Allergenic Extract | Placebo (Glycero-Cocas)
Number analyzed (Participants) | 192 | 192
Scores on a scale | 1.374 (2.10) | 2.231 (3.20)
Statistical Analysis 1: Comparison: Ragweed Allergenic Extract vs Placebo (Glycero-Cocas); Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = -0.857, 95% CI 2-sided [-1.388 to -0.326]

3. Secondary Outcome: Scores of a Scale (Average Daily Rhinoconjunctivitis Symptom Scores During the Entire Ragweed Pollen Season)
Description: Change in baseline in avg daily RSS during entire ragweed season in ITT population. Symptom score: sum of scores from 8 symptoms rated 0-3 (0=absent, 1=mild, 2=moderate, 3=severe), ocular (itchiness, swelling/redness, and watery eyes/tears), nasal (sneezing, itching, runny and stuffy nose), and ears (itching). Avg daily RSS Total Score Range: 0 (min) - 48 (max); lower score was more favorable. Avg daily RSS computed by: (1) summing 8 individual allergy symptoms recorded in AM and PM; (2) forming daily RSS by summing AM and PM RSS for each day of ragweed season; (3) averaging daily RSS for entire ragweed season.
Time Frame: 2011 ragweed pollen season; 8/2011 - 10/2011
Population: ITT population includes subjects who had at least one post treatment efficacy measurement
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ragweed Allergenic Extract | Placebo (Glycero-Cocas)
Number analyzed (Participants) | 196 | 193
Scores on a scale | 0.830 (1.56) | 1.601 (2.29)
Statistical Analysis 1: Comparison: Ragweed Allergenic Extract vs Placebo (Glycero-Cocas); Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = -0.771, 95% CI 2-sided [-1.213 to -0.329]

4. Secondary Outcome: Scores on a Scale (Average Daily Rhinoconjunctivitis Symptom Scores During the Three Peak Weeks of Ragweed Pollen Season)
Description: Change from baseline in avg daily rhinoconjunctivitis symptom scores during the three peak weeks of ragweed pollen season for the ITT population (netpRSS).
  Symptom score: sum of scores from 8 symptoms rated 0-3 (0=absent, 1=mild, 2=moderate, 3=severe), ocular (itchiness, swelling/redness, and watery eyes/tears), nasal (sneezing, itching, runny and stuffy nose), and ears (itching). Avg daily RSS Total Score Range: 0 (min) - 48 (max); lower score was more favorable. Avg daily RSS computed by: (1) summing 8 individual allergy symptoms recorded in AM and PM; (2) forming daily RSS by summing AM and PM RSS for each day of ragweed season; (3) averaging daily RSS for three peak weeks of ragweed pollen season.
Time Frame: 3 peak weeks of the 2011 ragweed pollen season
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Ragweed Allergenic Extract: Allergy Immunotherapy: Daily administration of Short Ragweed Allergenic Extract up to 42 U Amb a 1 for a minimum of 8 weeks prior to the ragweed pollen season.
  Short Ragweed Allergenic Extract: Active-Short Ragweed Allergenic Extract sublingual
Arm/Group | Ragweed Allergenic Extract | Placebo (Glycero-Cocas)
Number analyzed (Participants) | 192 | 192
Scores on a scale | 1.318 (1.99) | 2.105 (3.01)
Statistical Analysis 1: Comparison: Ragweed Allergenic Extract vs Placebo (Glycero-Cocas); Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = -0.788, 95% CI 2-sided [-1.291 to -0.284]

ADVERSE EVENTS:
Groups:
- Ragweed Allergenic Extract: allergy immunotherapy: Daily administration of ragweed allergenic extract up to 42U Amb a 1 for a minimum of 8 week prior to the ragweed pollen season.
  placebo and short ragweed allergenic extract: Active- short ragweed allergenic extract sublingual Placebo-Glycero-Cocas sublingual
- Glycero-Cocas: placebo and short ragweed allergenic extract: Active- short ragweed allergenic extract sublingual Placebo-Glycero-Cocas sublingual
Arm/Group | Ragweed Allergenic Extract | Glycero-Cocas
Serious Adverse Events (participants affected / at risk) | 2/218 | 3/211
Other Adverse Events (participants affected / at risk) | 28/218 | 29/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ragweed Allergenic Extract (N=218) | Glycero-Cocas (N=211)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ragweed Allergenic Extract (N=218) | Glycero-Cocas (N=211)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (11) | 22 (22)
Headache (Nervous system disorders) | 17 (17) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less